CLINICAL TRIAL: NCT05290974
Title: Comparison Between Self-directed Online Educational Material and Conventional Teaching in Acquiring Ultrasound-guided Regional Anesthesia Skills for Supraclavicular Brachial Plexus Block by Novice Performers
Brief Title: Online Regional Anesthesia Resources - Are They Effective?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, PGME Learner - Clinical Fellow, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MSH REB 22-0007-E
Record Dates: First submitted 2022-03-13; First posted 2022-03-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Education
Keywords: Regional Anesthesia; Ultrasonic Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person group (Active Comparator): Conventional in-person standardized teaching
  Interventions: Other: Conventional in-person teaching on supraclavicular brachial plexus block
- Online group (Experimental): Independent learning with online educational material
  Interventions: Other: Self exploring of available online material on supraclavicular brachial plexus block

INTERVENTIONS:
Other: Self exploring of available online material on supraclavicular brachial plexus block — Potential new method of learning a specific regional anesthesia technique
  Arms: Online group
Other: Conventional in-person teaching on supraclavicular brachial plexus block — Conventional method of learning a specific regional anesthesia technique
  Arms: In-person group

SUMMARY:
Anatomical-based ultrasound imaging has been one of the most rapidly advancing innovations in the field of regional anesthesia in recent years. The proper performance of ultrasound guided regional anesthesia (UGRA) is a useful competency for any anesthesiologist. However, there are some obstacles in regional anesthesia education for trainees. The increasing availability of UGRA related online information may have an important educational value for trainees and consultants. The objective of this study is to assess the impact of using educational material from The New York School of Regional Anesthesia (NYSORA) and Ultrasound for Regional Anesthesia (USRA) websites on image acquisition and anatomical interpretation learning process of novice trainees residents performing ultrasound guided supraclavicular brachial plexus block. We hypothesize that the use of those online educational materials will give learners non inferior ability and knowledge for image acquisition and anatomical interpretation of ultrasound image for supraclavicular brachial plexus block, when compared to conventional in person teaching.

DETAILED DESCRIPTION:
Introduction Anatomical-based ultrasound imaging has been one of the most rapidly advancing innovations in the field of regional anesthesia in recent years. Compared with landmark based or peripheral nerve stimulation techniques, benefits of ultrasound guided regional anesthesia (UGRA) include increased nerve block success rate, faster onset time, decreased volume of local anesthetic, and reduced risk of complications. Most experts now consider ultrasound-guidance to be the standard of care for peripheral nerve blocks. To successfully perform a UGRA procedure, a triad of three distinct but interrelated skills is required: image acquisition and anatomical interpretation are needed to identify the needle insertion point; hand-eye coordination is then needed to advance the needle to the target. First, the clinician must successfully acquire an image and then correctly interpret the sonoanatomy. Next, the needle must be visualized and guided to the desired target. This dynamic process often requires constant needle manipulation with simultaneous adjustments of the ultrasound transducer.

The proper performance of UGRA is a useful competency for any anesthesiologist, and most anesthesia residency programs are required to have a minimum curriculum for education of the most frequent and well stablished peripheral nerve blocks. However, there are some obstacles in regional anesthesia education for trainees. The traditional "apprenticeship model" of learning while concurrently providing clinical care can result in inconsistent learning experiences, variability in case numbers, and compromised patient safety. It is not feasible to practice all UGRA steps (especially needling) in live voluntary models. Simulation-based techniques (animal, cadavers) can be expensive and logistically difficult to use on a regular basis. Conventional regional anesthesia training in most regional anesthesia courses and workshops consists of theoretical teaching (in-person instruction of indications, anatomical concepts, techniques and complications) followed by hands-on image acquisition demonstration and practice on live voluntary models. This structured teaching method can be impractical in a medical residency program, where time constraints during clinical care can limit teaching opportunities. Moreover, for novices, it provides a brief, isolated exposure to the procedure, which limits long-term retention and associated with decay of skill execution.

There is a growing availability of online UGRA related material, including good quality open access educational information, assembled by related societies (The New York School of Regional Anesthesia - NYSORA; Ultrasound for Regional Anesthesia - USRA). Therefore, an opportunity may exist for using this kind of content for UGRA learning in anesthesiology medical residency programs.

Significance The increasing availability of UGRA related online information may have an important educational value for trainees and consultants. The structured use of this material, can contribute to learners' skill acquisition and reduce requirements for human resources and time needed for UGRA training. It also provides easy access to review skills to improve retain competency.

Objectives To assess the impact of using educational material from NYSORA and USRA websites on image acquisition and anatomical interpretation learning process of novice trainees performing supraclavicular brachial plexus block.

Hypothesis Use of online educational materials for ultrasound guided supraclavicular brachial plexus from NYSORA and USRA will give learners non inferior ability and knowledge for image acquisition and anatomical interpretation of ultrasound image for supraclavicular brachial plexus block, when compared to conventional in person teaching.

Methods Study type Single-center randomized controlled trial, blinded for evaluator, comparing two educational strategies (directed independent learning with online educational material versus conventional in-person teaching) in acquiring two ultrasound-guided regional anesthesia skills (image acquisition and anatomical interpretation) for supraclavicular brachial plexus block, among novice to UGRA (University of Toronto first year anesthesiology residents, rotating at Sinai Health System - Mount Sinai Hospital). Following Ethics Research Board approval, subjects will be recruited for the study. Their eligibility for participation will be assessed and they will be consented for voluntary participation in the study by signing an informed written consent.

Study interventions The participants will be randomized to one of the two groups using a computer-generated random numbers table: in-person standardized teaching group (in-person group) or independent learning with online educational material group (online group).

The participants randomized to the in-person group will be scheduled for a standardized in-person theoretical teaching session, performed by the same anesthesiologist with wide experience in ultrasound guided supraclavicular brachial plexus block. The in-person teaching will involve a maximum of five learners per session.

The online group will not participate in any in-person teaching. This group will receive the online material for self-directed reading and exploration (including available figures and videos). The educational material from NYSORA (available on: https://www.nysora.com/regional-anesthesia-for-specific-surgical-procedures/upper-extremity-regional-anesthesia-for-specific-surgical-procedures/anesthesia-and-analgesia-for-elbow-and-forearm-procedures/ultrasound-guided-supraclavicular-brachial-plexus-block/) and USRA (available on: http://www.usra.ca/regional-anesthesia/specific-blocks/upper-limb/suprablock.php) websites are going to be used, and were selected because of their high quality, validated in other studies. It is not possible to ensure the in-person group does not also utilize online resources in preparation, a key factor will be explicit direction to the online group to review these specific high-quality resources.

All participants will be requested to be present for a practical demonstration of ultrasound imaging acquisition and skill evaluation, within two weeks following the in-person teaching or online material independent learning. Participants will demonstrate the technique they will have learned, in the same live model volunteer for both groups. They will use the same equipment (Edge II; Sonosite, Bothel, Washington.). They will try to acquire the best ultrasound image for an optimal ultrasound guided right supraclavicular brachial plexus block, under evaluation of the same UGRA experienced evaluator. Participants' performance will be evaluated using a checklist for acquiring and interpreting the sonogram of key neural and nonneural structures relevant to ultrasound guided supraclavicular brachial plexus block. This checklist was adapted from previous studies [appendix 1 - Sonographic Proficiency Assessment Score (SPAS) for Supraclavicular Brachial Plexus Block]. It generates a score that ranges from 0 to 33. This checklist assesses participants' performance based on their capability to describe and demonstrate the indications of the block; territorial distribution of anesthesia; patient position; range of sterility; correct transducer option and position; anatomical structures on ultrasound image; needle insertion; direction and final position; expected local anesthetic spread; adequate local anesthetic volume; possible complications and how to avoid them. The evaluator for participants' SPAS will be blinded for which group they were randomized to. The best acquired image demonstrating the required landmarks will also be captured and later assessed by an independent blinded evaluator.

Sample size There is no previous data in the literature comparing the independent use of online educational material with conventional in person teaching, for image acquisition and anatomical interpretation of ultrasound image for supraclavicular brachial plexus block. Sample size was therefore based on a previous study comparing the effect of two methods on the learning curve for acquiring sonographic skills for axillary brachial plexus block, among ten medical students. In order to achieve a larger power than the aforementioned study, recruitment and randomization of 20 PGY1s is planned..

Study data analysis Normal distributed variables values will be presented and analyzed as mean values +- standard deviation. Non-normal distributed variables values will be presented and analyzed as median and minimum and maximum values. Qualitative variables will be presented as frequency of occurrence. Statistical test to be performed might be: t-Student, Kruskal-Wallis and Chi-square. Statistical software will be used for analysis: SPSS 13.0 for Windows (SPSS Inc, Chicago, IL, USA) and GraphPad Prism Version 4.00 for Windows (GraphPad Software, San Diego, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* First year anesthesiology residents, willing to be present for a standardized in-person teaching module or perform an independent study of standardized online material, with no more than one previously performed supraclavicular ultrasound guided block, and willing to undergo to an anonymous skill acquisition assessment.

Exclusion Criteria:

* Learner refusal to participate and decision to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Sonographic Proficiency Assessment Score for Supraclavicular Brachial Plexus Block | Two weeks
  Checklist for acquiring and interpreting the sonogram of key neural and nonneural structures relevant to ultrasound guided supraclavicular brachial plexus block

SECONDARY OUTCOMES:
Quality of the acquired image | Two weeks
  Quality of the best acquired image by two experienced anesthesiologists

CONTACTS AND LOCATIONS:
Overall Officials: Hermann dos Santos Fernandes, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Make individual anonymized data available, after the conclusion of the study, through a RedCap exported data sheet.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study on scientific journal.

REFERENCES:
- [Background] Barrington MJ, Kluger R. Ultrasound guidance reduces the risk of local anesthetic systemic toxicity following peripheral nerve blockade. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):289-99. doi: 10.1097/AAP.0b013e318292669b. PMID 23788067
- [Background] Marhofer P, Harrop-Griffiths W, Kettner SC, Kirchmair L. Fifteen years of ultrasound guidance in regional anaesthesia: part 1. Br J Anaesth. 2010 May;104(5):538-46. doi: 10.1093/bja/aeq069. Epub 2010 Apr 2. PMID 20364022
- [Background] Chen XX, Trivedi V, AlSaflan AA, Todd SC, Tricco AC, McCartney CJL, Boet S. Ultrasound-Guided Regional Anesthesia Simulation Training: A Systematic Review. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):741-750. doi: 10.1097/AAP.0000000000000639. PMID 28759501
- [Background] Kim TE, Tsui BCH. Simulation-based ultrasound-guided regional anesthesia curriculum for anesthesiology residents. Korean J Anesthesiol. 2019 Feb;72(1):13-23. doi: 10.4097/kja.d.18.00317. Epub 2018 Nov 27. PMID 30481945
- [Background] Smith HM, Kopp SL, Jacob AK, Torsher LC, Hebl JR. Designing and implementing a comprehensive learner-centered regional anesthesia curriculum. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):88-94. doi: 10.1097/AAP.0b013e31819e734f. No abstract available. PMID 19282705
- [Background] Ramirez AG, Hu Y, Kim H, Rasmussen SK. Long-Term Skills Retention Following a Randomized Prospective Trial on Adaptive Procedural Training. J Surg Educ. 2018 Nov;75(6):1589-1597. doi: 10.1016/j.jsurg.2018.03.007. Epub 2018 May 24. PMID 29803772
- [Background] Tewfik GL, Work AN, Shulman SM, Discepola P. Objective validation of YouTube educational videos for the instruction of regional anesthesia nerve blocks: a novel approach. BMC Anesthesiol. 2020 Jul 9;20(1):168. doi: 10.1186/s12871-020-01084-w. PMID 32646371
- [Background] Barrington MJ, Viero LP, Kluger R, Clarke AL, Ivanusic JJ, Wong DM. Determining the Learning Curve for Acquiring Core Sonographic Skills for Ultrasound-Guided Axillary Brachial Plexus Block. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):667-670. doi: 10.1097/AAP.0000000000000487. PMID 27685348
- [Background] Udani AD, Harrison TK, Mariano ER, Derby R, Kan J, Ganaway T, Shum C, Gaba DM, Tanaka P, Kou A, Howard SK; ADAPT (Anesthesiology-Directed Advanced Procedural Training) Research Group. Comparative-Effectiveness of Simulation-Based Deliberate Practice Versus Self-Guided Practice on Resident Anesthesiologists' Acquisition of Ultrasound-Guided Regional Anesthesia Skills. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):151-7. doi: 10.1097/AAP.0000000000000361. PMID 26866296